CLINICAL TRIAL: NCT03963817
Title: Snapshot 3D Ultra-high-resolution OCT and Hyperspectral AF of In-vivo Retina
Brief Title: Snapshot Camera for AMD
Status: Active, not recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of California, Los Angeles (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Roland Theodore Smith, MD, PhD, Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 17-1999; 1R01EY029397-01A1 (NIH)
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Age Related Macular Degeneration
Keywords: Imaging; Autofluorescence imaging; Spectral domain optical coherence tomography; Adaptive optics; Soft drusen; Reticular pseudodrusen
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normals: Imaging normal subjects for equipment refinement
  Interventions: Diagnostic Test: adaptive optics AO-OCT/AF instrument
- Subjects with AMD: Imaging subjects with AMD
  Interventions: Diagnostic Test: adaptive optics AO-OCT/AF instrument

INTERVENTIONS:
Diagnostic Test: adaptive optics AO-OCT/AF instrument — Using the new adaptive optics AO-OCT/AF instrument, the study team will image 10 normal subjects in order to optimize image acquisition and interpretation.
  Other Names: Normals
  Groups: Normals
Diagnostic Test: adaptive optics AO-OCT/AF instrument — Using the new adaptive optics AO-OCT/AF instrument, the study team will image 40 adult subjects with age-related macular degeneration (AMD) who have non-neovascular AMD and soft drusen or subretinal drusenoid deposits in the macula.
  Other Names: AMD
  Groups: Subjects with AMD

SUMMARY:
This study proposes to use a new instrument (AO-OCT/AF: adaptive optics - optical coherence tomography/autofluorescence) combined with a data processing method to image the retinal pigment epithelium (RPE) of the eye in normal subjects and in subjects with age-related macular degeneration. (AMD). While currently there is no cure, with early diagnosis, vision loss can be slowed. The technology being developed for this project will be the first imaging modality that can provide both structural and molecular information about the retina in vivo and in 3D.

DETAILED DESCRIPTION:
An imaging modality that allows for fast, simultaneous, noninvasive probing of both 3D cellular resolution retinal morphology by optical coherence tomography (OCT) and molecular-specific functions by autofluorescence (AF) could substantially improve both basic understanding and the early diagnosis of age-related macular degeneration (AMD), the leading cause of blindness in the developed world. The evaluation and management of AMD utilize several investigation modalities, but advancements in OCT technology have significantly contributed to better understanding of the disease, and have helped with monitoring progression and therapeutic efficacy. However, due to optical aberrations of the eye, the transverse resolution of conventional OCT is generally limited to 10-15 µm, restricting its use to visualize individual retinal cells in vivo. The integration of adaptive optics (AO) into OCT has demonstrated an immense success in mitigating these aberrations. Among various AO-OCT techniques, computation-based AO (CAO) becomes the spotlight of research because it shows unique advantages in data postprocessing flexibility and a reduced system cost. However, CAO is extremely sensitive to phase stability. The rapid motion of the eye can easily scramble the phase of reflected photons, restricting imaging to a single en-face layer.

To overcome this problem, the study team will integrate a snapshot hyperspectral imaging method, Image Mapping Spectrometry (IMS), with full-field spectral-domain OCT. The integrated system will first enable 3D CAO imaging of the retina because the single camera exposure (4 s),is too fast for eye movement to scramble phase between layers. Next, to improve resolution in 3D, the study team will adapt an established CAO algorithm to correct for wavefront aberrations. The resultant method, which the study team terms snapshot ultra-high-resolution OCT, will allow an acquisition of a quarter million A-scans simultaneously. Given a typical flash illumination duration (4us), the equivalent A-scan rate is 62.5 GHz, which is approximately three orders of magnitude faster than the state-of-the-art methods. Furthermore, to expand the system's functionality to molecular imaging, the study team will add a second IMS imaging channel for simultaneous hyperspectral imaging of retinal pigment epithelium (RPE) AF, enabling spectral biopsy of RPE and subRPE lesions such as drusen, the hallmark lesion of early AMD. The resultant dual-channel AO-OCT/AF system will be the first imaging modality that can provide both structural and molecular information about the retina in vivo and in 3D. The study team envisions such a system would shift the landscape of AMD evaluation and management. The insights so obtained will be of high value in clinical diagnosis and treatment. In addition, such a system will accelerate translational research with sensitive and early outcome testing of prospective therapeutic agents, saving sight and thereby providing enormous benefit to society.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged 60 and over and pseudophakic, with clear posterior capsule and dilation to 6mm.
* Patients must be diagnosed early/intermediate AMD in at least one eye (the study eye) with soft drusen or reticular pseudodrusen in the macula.

Exclusion Criteria:

* Retinopathy other than AMD.
* Inability to give informed consent
* Bilateral advanced AMD
* Allergy to dilation eye drops

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from referring physicians of the faculty practice of New York Eye and Ear Infirmary of Mount Sinai
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Excitation spectra | 3 years
  Excitation spectra of the retinal tissue at or near 436 nm, which will be considered representative of drusen or drusenoid material

SECONDARY OUTCOMES:
Emission spectra | 3 years
  Emission spectra of the retinal tissue at or near 510 nm, which will be considered representative of drusen or drusenoid material

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Theodore Smith, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- New York Eye and Ear Infirmary of Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Results of the study will be shared as publications in peer-reviewed journals and at scientific meetings.